CLINICAL TRIAL: NCT02400437
Title: Phase II Trial of Ixazomib, Dexamethasone and Rituximab in Patients With Untreated Waldenstrom's Macroglobulinemia
Brief Title: Trial of Ixazomib, Dexamethasone and Rituximab in Patients With Untreated Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Jorge J. Castillo, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-559
Record Dates: First submitted 2015-03-10; First posted 2015-03-27 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: Waldenstrom's Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — ixazomib; Dexamethasone; Calcium Dobesilate; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IDR (Experimental): - IDR The study treatment will consist on an induction and a maintenance phase. Dose modification will be permitted for toxicity
  * Induction cycles will be 4 weeks long, Maintenance cycles 8 weeks long.
  * Ixazomib- administered orally on predetermined days and dosage during Induction and Maintenance Phase
  * Dexamethasone- administered via IV or orally on predetermined days and dosage during Induction and Maintenance Phase
  * Rituximab- administered via IV on predetermined days and dosage during Induction and Maintenance Phase
  Interventions: Drug: Ixazomib; Drug: Dexamethasone; Drug: Rituximab

INTERVENTIONS:
Drug: Ixazomib — Doses given on Days 1, 8, and 15 in induction and maintenance cycles.
  Other Names: MLN9708
Drug: Dexamethasone — Doses given on Days 1, 8, and 15 in induction and maintenance cycles.
  Other Names: Decadron; Dexasone,; Diodex; Hexadrol; Maxidex
Drug: Rituximab — Doses given on Day 1 of induction and maintenance cycles.
  Other Names: Rituxan

SUMMARY:
This research study is evaluating a drug called ixazomib (also known as MLN9708) in combination with dexamethasone and rituximab (the regimen is called IDR) as a possible treatment for Waldenstrom's Macroglobulinemia (WM).

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational regimen, IDR, to learn whether IDR works in treating a specific cancer. "Investigational" means that IDR is still being studied and that research doctors are trying to find out more about it-such as the safest dose to use, the side effects it may cause, and if IDR is effective for treating different types of cancer. It also means that the FDA (the U.S. Food and Drug Administration) has not yet approved IDR for use in participants with your type of cancer.

Ixazomib is a drug that may kill or stop cancer cells from growing by blocking the proteasome within the cell, which is responsible for degrading or breaking down a variety of proteins. This type of drug is called a proteasome inhibitor.

Rituximab is a type of protein called an antibody that attacks the cluster of differentiation 20 (CD20), a protein found on B-cells like WM. Rituximab is approved by the FDA for treating non-Hodgkin lymphoma (NHL). Dexamethasone is a steroid and is similar to the hormones naturally produced by the adrenal glands; it prevents the release of substances that cause inflammation. Rituximab and dexamethasone are often used to treat WM, alone or in combination with other drugs. Combinations with rituximab, dexamethasone and other proteasome inhibitors have shown good response rates in WM participants. Ixazomib is a proteasome inhibitor; thus the investigator swill investigate if the combination of Ixazomib, Rituximab, and Dexamethasone is also active in WM.

In this research study, the investigators are combining a new treatment ixazomib with a standard regimen, rituximab and dexamethasone, to determine whether this combination (IDR) is effective and safe for participants with previously untreated WM.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older.
* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that the patient may withdraw consent at any time without prejudice to future medical care.
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Clinicopathological diagnosis of WM (Owen 2003), with symptomatic disease meeting criteria for treatment using consensus panel criteria from the Second International Workshop on WM (Kyle 2003), and measurable disease, defined as presence of immunoglobulin M (IgM) paraprotein with a minimum IgM level of >2 times the upper limit of normal.
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2.
* Patients must meet the following clinical laboratory criteria
* Absolute neutrophil count ≥1,000/mm3 and platelet count ≥75,000/mm3. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.
* Total bilirubin ≤1.5 x the upper limit of the normal range (ULN).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x ULN.
* Calculated creatinine clearance ≥30 mL/min.

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period.
* Major surgery within 14 days before enrollment.
* Central nervous system involvement.
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Systemic treatment, within 14 days before the first dose, with strong inhibitors of cytochrome P (CYP) 1A2, strong inhibitors of CYP3A, or strong CYP3A inducers, or use of Ginkgo biloba or St. John's wort.
* Known hepatitis B or C virus, or HIV infection.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-04; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge J. Castillo, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Castillo JJ, Meid K, Flynn CA, Chen J, Demos MG, Guerrera ML, Kofides A, Liu X, Munshi M, Tsakmaklis N, Patterson CJ, Yang G, Hunter Z, Treon SP. Ixazomib, dexamethasone, and rituximab in treatment-naive patients with Waldenstrom macroglobulinemia: long-term follow-up. Blood Adv. 2020 Aug 25;4(16):3952-3959. doi: 10.1182/bloodadvances.2020001963. PMID 32822482
- [Derived] Castillo JJ, Meid K, Gustine JN, Dubeau T, Severns P, Hunter ZR, Yang G, Xu L, Treon SP. Prospective Clinical Trial of Ixazomib, Dexamethasone, and Rituximab as Primary Therapy in Waldenstrom Macroglobulinemia. Clin Cancer Res. 2018 Jul 15;24(14):3247-3252. doi: 10.1158/1078-0432.CCR-18-0152. Epub 2018 Apr 16. PMID 29661775

RESULTS

PARTICIPANT FLOW:
Groups:
- Ixazomib, Dexamethasone, Rituximab: - IDR The study treatment will consist on an induction and a maintenance phase. Dose modification will be permitted for toxicity
  * Induction cycles will be 4 weeks long, Maintenance cycles 8 weeks long.
  * Ixazomib- administered orally on predetermined days and dosage during Induction and Maintenance Phase
  * Dexamethasone- administered via IV or orally on predetermined days and dosage during Induction and Maintenance Phase
  * Rituximab- administered via IV on predetermined days and dosage during Induction and Maintenance Phase
  Ixazomib: Doses given on Days 1, 8, and 15 in induction and maintenance cycles.
  Dexamethasone: Doses given on Days 1, 8, and 15 in induction and maintenance cycles.
  Rituximab: Doses given on Day 1 of induction and maintenance cycles.
Period: Overall Study
Arm/Group | Ixazomib, Dexamethasone, Rituximab
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants are included in the analysis.
Arm/Group | Ixazomib, Dexamethasone, Rituximab
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 15
Age, Continuous [Median (Full Range); unit: years] | 62.5 [46 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26
Mutational Status [Count of Participants; unit: Participants]
  MYD88 Mutated, CXCR4 Wild-type | 11
  MYD88 Mutated, CXCR4 Mutated | 15

OUTCOME MEASURES:

1. Primary Outcome: Very Good Partial Response Rate (VGPR) for IDR
Description: Rate of very good partial response or better in patients treated with IDR. VGPR is defined as a >90% reduction in serum IgM levels from baseline.
Time Frame: 76 weeks
Population: All participants who have received at least 1 cycle of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib, Dexamethasone, Rituximab
Number analyzed (Participants) | 26
Participants | 5

2. Secondary Outcome: Overall Response Rate
Description: Overall response includes the rate of complete response (CR), partial response (PR), minimal response (MR), stabl disease (SD) and progressive disease (PD). Minor response is >25%-50% reduction in serum IgM from baseline. Partial Response is (>50-90% reduction in serum IgM from baseline. Very Good Partial Response is >90% reduction in serum IgM from baseline. Complete Response is resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly.
Time Frame: 2 Years
Population: All participants who received at least 1 cycle of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib, Dexamethasone, Rituximab
Number analyzed (Participants) | 26
Participants | 25

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Duration of time from start of treatment to disease progression. Progressive disease is defined as occurring when a >25% increase in serum IgM and an absolute 500mg/dL increase in IgM level occurs from the lowest attained response value, or progression of clinically significant disease related symptoms.
Time Frame: From start of treatment to time of disease progression, assessed up to 4 years after treatment start
Population: All participants who received at least 1 cycle of therapy. Participants were followed for up to 2 years after treatment discontinuation.
Measure: Median (Full Range); unit: months
Arm/Group | Ixazomib, Dexamethasone, Rituximab
Number analyzed (Participants) | 26
months | 33 [4 to 46]

4. Secondary Outcome: Overall Response Rate by MYD88 L265P and CXCR4-WHIM Status
Description: To evaluate the overall response rate of participants by MYD88 L265P and CXCR4-WHIM mutations in WM. Overall response is defined as achieving at least a minor response, or >25% reduction in serum IgM from baseline.
Time Frame: 2 Years
Population: Number of participants who achieved a response by mutational status
Measure: Count of Participants; unit: Participants
Groups:
- MYD88 Mutated, CXCR4 Wild-type: Participants who were MYD88 mutated and did not have the CXCR4 mutation
- MYD88 Mutated, CXCR4 Mutated: Participants with both the MYD88 mutation and a CXCR4 mutation
Arm/Group | MYD88 Mutated, CXCR4 Wild-type | MYD88 Mutated, CXCR4 Mutated
Number analyzed (Participants) | 11 | 15
Participants | 11 | 14

5. Secondary Outcome: Time to Progression (TTP)
Description: Duration of time from start of treatment to time of disease progression.
Time Frame: From start of treatment to time of disease progression, assessed up to 4 years after treatment start
Population: All participants who received 1 cycle of treatment.
Measure: Median (Full Range); unit: months
Arm/Group | Ixazomib, Dexamethasone, Rituximab
Number analyzed (Participants) | 26
months | 33 [4 to 46]

6. Secondary Outcome: Duration of Response (DOR)
Description: The duration of response is measured from the time a participant achieved a response until the date of progression.
Time Frame: From the time each participant achieved a response to time of disease progression, assessed up to 4 years after treatment start
Population: All participants who achieved a response to therapy.
Measure: Median (Full Range); unit: months
Arm/Group | Ixazomib, Dexamethasone, Rituximab
Number analyzed (Participants) | 25
months | 33 [2 to 41]

7. Secondary Outcome: Time to Next Therapy (TTNT)
Description: Duration from start of protocol treatment to time of initiation of new therapy.
Time Frame: From start of treatment until the participant begins a new therapy, assessed up to 4 years after treatment start
Measure: Median (Full Range); unit: months
Arm/Group | Ixazomib, Dexamethasone, Rituximab
Number analyzed (Participants) | 26
months | 39 [4 to 46]

ADVERSE EVENTS:
Time Frame: Adverse events were collected starting after the first dose of study medication through 30 days of last treatment, an average of 1.5 years.
Arm/Group | Ixazomib, Dexamethasone, Rituximab
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 4/26
Other Adverse Events (participants affected / at risk) | 25/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixazomib, Dexamethasone, Rituximab (N=26)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Failure to thrive (General disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Flu-like symptoms (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Staph Aureus Bacteremia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixazomib, Dexamethasone, Rituximab (N=26)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Blurry vision (Eye disorders) | 3 (3)
Cataract (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (9)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4)
Chills (General disorders) | 4 (4)
Edema face (General disorders) | 3 (3)
Fatigue (General disorders) | 9 (9)
Fever (General disorders) | 6 (6)
Flu-like symptoms (General disorders) | 1 (1)
Feeling cold (General disorders) | 1 (1)
Sweats (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 9 (9)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 2 (2)
Unspecified rash (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 9 (9)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (6)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 2 (2)
Shoulder discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Thyroid nodules (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 6 (6)
Dysgeusia (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (7)
Presyncope (Nervous system disorders) | 1 (1)
Sinus pressure (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 8 (8)
Restless legs (Psychiatric disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Amenorrhea (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 5 (5)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Hematoma (Vascular disorders) | 2 (2)
Hot flashes (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT02400437/Prot_SAP_000.pdf